CLINICAL TRIAL: NCT00271557
Title: A Randomized, Open-Label, Active-Controlled, Multicenter Phase III Safety Study of Two Doses of NATRECOR hBNP (Nesiritide) Administered as a Continuous Infusion in the Treatment of Decompensated CHF
Brief Title: A Study to Develop Additional Safety and Clinical Experience With NATRECOR hBNP (Nesiritide) in the Treatment of Patients With Worsening Congestive Heart Failure Who Require Inpatient Intravenous Therapy With Medications That Influence the Tone and Caliber of Blood Vessels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005203
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Heart Failure, Congestive; Heart Decompensation
Keywords: Heart Failure; Renal Dysfunction; Cardiomyopathy; Heart Decompensation; Dyspnea Paroxysmal.
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardiomyopathies; Dyspnea, Paroxysmal | interventions — Natriuretic Peptide, Brain

INTERVENTIONS:
Drug: nesiritide

SUMMARY:
The purpose of this safety study is to evaluate NATRECORÂ® hBNP (a recombinant form of the natural human peptide normally secreted by the heart in response to heart failure), in subjects with worsening congestive heart failure for whom inpatient intravenous therapy with medications that influence the tone and caliber of blood vessels is deemed appropriate.

DETAILED DESCRIPTION:
The data from these previous studies suggest that doses of NATRECOR® hBNP may be a potent agent for the treatment of acute congestive heart failure (CHF) with a unique combination of desirable effects on the flow of blood throughout the body; the hormones secreted by the nervous system; and support of copious salt outputs by the renal system not provided by currently available therapies. The purpose of this safety study is to evaluate NATRECOR® hBNP in subjects with symptomatic, decompensated congestive heart failure for whom inpatient intravenous therapy with medications that influence the tone and caliber of blood vessels (other than, or in addition to, IV diuretics) is deemed appropriate. This is a multi-center, randomized, open-label, safety study designed to compare two doses of NATRECOR® hBNP for the treatment of decompensated congestive heart failure. One treatment group receives NATRECOR® hBNP fixed-dose infusion IV bolus of 0.3 µg/kg followed by a 0.015 µg/kg/min infusion; group two receives IV bolus of 0.6 µg/kg followed by a 0.03 µg/kg/min infusion. The duration of NATRECOR® hBNP therapy is determined by the attending physician. The study hypothesis is that doses of NATRECOR® hBNP in the range of 0.015 to 0.03 µg/kg/min provide an optimal safety/efficacy profile for the treatment of decompensated CHF. One treatment group receives NATRECOR® hBNP fixed-dose infusion IV bolus of 0.3 µg/kg followed by a 0.015 µg/kg/min infusion; group two receives IV bolus of 0.6 µg/kg followed by a 0.03 µg/kg/min infusion. The duration of NATRECOR® hBNP therapy is determined by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous history of chronic congestive heart failure (CHF)
* presenting with symptomatic, decompensated CHF for inpatient intravenous therapy with medications that influence the tone and caliber of blood vessels (other than, or in addition to, diuretics)

Exclusion Criteria:

* Patients with myocardial ischemia within the past 48 hours
* having significant valvular stenosis, obstructive cardiomyopathy, constrictive pericarditis or primary pulmonary hypertension
* being treated with intravenous (IV) therapy with medications that influence the tone and caliber of blood vessels for > 4 hours for this episode of CHF
* already being treated with IV therapy with medications that influence the tone and caliber of blood vessels that cannot be discontinued
* having cardiogenic shock, systolic blood pressure consistently < 90 mm Hg or other significant blood circulation instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 1997-01; Study Completion 1997-12 (Actual)

PRIMARY OUTCOMES:
Changes in symptoms and signs of CHF after 6 hours and after 24 hours of treatment with NATRECOR® hBNP.

SECONDARY OUTCOMES:
Adverse events, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Result] Mills RM, LeJemtel TH, Horton DP, Liang C, Lang R, Silver MA, Lui C, Chatterjee K. Sustained hemodynamic effects of an infusion of nesiritide (human b-type natriuretic peptide) in heart failure: a randomized, double-blind, placebo-controlled clinical trial. Natrecor Study Group. J Am Coll Cardiol. 1999 Jul;34(1):155-62. doi: 10.1016/s0735-1097(99)00184-9. PMID 10400005